CLINICAL TRIAL: NCT01270477
Title: Study of the Possible Improvement in Level of Sequela and Amputation/Amputation Level After Frost Injury by the Adjuvant Treatment of Hyperbaric Oxygen.
Brief Title: Hyperbaric Oxygen Treatment as Adjuvant Treatment for Frost Injury
Acronym: FROST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of People to follow up the study, work overload
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Helle Midtgaard, Physiscian, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FROST
Record Dates: First submitted 2011-01-03; First posted 2011-01-05 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2011-04

CONDITIONS: Wound (Morphologic Abnormality)
Keywords: Frost injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen treatment (Experimental): Hyperbaric oxygen treatment in an hyperbaric oxygen treatment chamber on an recognized treatment table.
  Interventions: Other: Hyperbaric oxygen treatment

INTERVENTIONS:
Other: Hyperbaric oxygen treatment — Hyperbaric oxygen treatment for 2,5 hours at maximum 14 meters (standard table in Norway).
  Other Names: Hyperoxic treatment; Pressure chamber treatment

SUMMARY:
The aim of this study is to see weather hyperbaric oxygen treatment is beneficial as adjuvant treatment for frost damage.

The investigators hope to include at least 20 patients in a randomized manner. Half of the patients are randomized to hyperbaric oxygen, and half of the patients are randomized not to have hyperbaric oxygen treatment.

Under hypotheses: The number og surgeries is reduced by hyperbaric oxygen treatment as adjuvant treatment for frost damage. The functional level of the frost damaged patient is better after 6 and 12 months when also treated with hyperbaric oxygen treatment for frost damage.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70. Frost damage grade II-IV. Inclusion is needed within 48 hours from time of damage.

Exclusion Criteria:

* Pregnancy. Ventilator treatment. Problems with equalizing. High grade heart failure. Chronic obstructive lung disease of high grade. Treatment over 3 days after time of damage. Serious claustrophobia/psychiatric illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-01; Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

PRIMARY OUTCOMES:
Hyperbaric oxygen treatment is favorable for tissue regeneration after frost injury. | From incusion of a patiant through a follow up after 1 year.

SECONDARY OUTCOMES:
First: The number of surgeries is reduced with hyperbaric oxygen treatment. | One year from the enrollment of a patient.
  Second: The level of amputation is further distal on the extremity with hyperbaric oxygen treatment.
  Third: The level of function of the damaged bodypart is better after 6 and 12 months with hyperbaric treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Knut Ar Kirkeboen, MD Professor, Study Director — Oslo University Hospital
Locations (1):
- Hyperbaric section Oslo University hospital, Oslo, Norway